CLINICAL TRIAL: NCT05979753
Title: Effects Of High Intensity Interval Training On Speed And Explosive Strength In Sprinters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Riphah123
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Sprinters

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFFECTS OF HIGH INTENSITY INTERVAL TRAINING IN SPRINTERS (Active Comparator): The aim of this is study is to assess the effect of High Intensity Interval Training on Sprinter's speed and explosive strength.
  Interventions: Other: EFFECTS OF HIGH INTENSITY INTERVAL TRAINING IN SPRINTERS
- EFFECTS OF HIGH INTENSITY INTERVAL TRAINING ON SPEED AND EXPLOSIVE STRENGTH (Active Comparator): The aim of this is study is to assess the effect of High Intensity Interval Training on Sprinter's speed and explosive strength.
  Interventions: Other: EFFECTS OF HIGH INTENSITY INTERVAL TRAINING IN SPRINTERS

INTERVENTIONS:
Other: EFFECTS OF HIGH INTENSITY INTERVAL TRAINING IN SPRINTERS — EFFECTS OF HIGH INTENSITY INTERVAL TRAINING ON SPEED AND EXPLOSIVE STRENGTH IN SPRINTER

SUMMARY:
High Intensity Interval Training (HIIT) is a type of exercise that alternates between short bursts of high and low intensity activity. The physical components may be improved very effectively and efficiently with this kind of training. The choice of an effective practice strategy could be very beneficial because boosting an athlete's performance is correlated with improving their physical components. The significance of this study was that HIIT is helpful in increasing strength, endurance and agility. Thus it could be useful for athletes for their physical fitness in less duration as compared to the conventional protocols.

DETAILED DESCRIPTION:
According to researchers knowledge there is lack of sufficient literature on "The Effect Of High Interval Intensity Training On Speed And Explosive Strength In Sprinters." The past trials do not address speed and strength in relation to HIIT and this study will help identify the need to practice this training in order to enhance the skills and athletic performance of sprinters and will uplift their anaerobic fitness.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 to 30 years
* Actively competing in races
* Had professional sprinting experience of one year
* Both genders included.
* Athletes who have clean bill of health for past 6 months
* Never engaged in a high intensity training program

Exclusion Criteria:

* Any Neuromuscular issue like myopathy, peripheral neuropathy and multiple sclerosis
* Any Musculoskeletal issue like chronic low back pain, tendinopathies, disc slips and OA
* Pregnancy
* Athlete who is on any kind of medications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
High Intensity Interval Training | 6 Months
  It consists of athletes who will perform these exercises 4 sessions per week for the period of 5 weeks.
  * 100 m runs with 30 seconds rest
  * 400 m runs with 90 seconds rest
  * Bouts of 120 second runs with 120 second rest
  * 30 second all out running sprinting with 3-minute rest
  * Duration and intensity of exercises will be modified accordingly
Conventional Exercises | 6 Months
  In this group athletes will perform conventional exercises as follows:
  * Squats.
  * Step Ups.
  * Deadlifts.
  * Heavy Sled Pulls.
  * Leg Press.
  * Single Leg Calf Extensions.
  * Jump Squats.
  * Bodyweight Jumps

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Shafique, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No